CLINICAL TRIAL: NCT05101590
Title: A Study of the Use, Safety and Efficacy of the Hypotension Decision Assist Device
Brief Title: Hypotension Decision Assist - Use, Safety and Efficacy
Acronym: HDA-USE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Directed Systems Limited (Industry)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BPA-CIP-001
Record Dates: First submitted 2021-10-01; First posted 2021-11-01 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Intraoperative Hypotension
Keywords: Hypotension; Intraoperative care; Intraoperative complications
MeSH Terms: conditions — Hypotension; Intraoperative Complications

STUDY DESIGN:
Intervention Model Description: Monitored with HDA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitored with HDA (Experimental): Participants undergoing elective major surgery and have an arterial line as part of their standard care with HDA included as part of their care
  Interventions: Device: Monitored by HDA

INTERVENTIONS:
Device: Monitored by HDA — Participants undergoing elective major surgery with an arterial line as part of their standard care and additional monitoring with HDA as part of their care.

SUMMARY:
This clinical investigation will investigate whether Hypotension Decision Assist (HDA) is a feasible, safe and effective patient clinical decision support system to enhance an anaesthetist's ability to manage a patient's cardiovascular system when undergoing surgery. If successful, this study will provide evidence that the use of HDA facilitates beneficial outcomes for patients who have this device used.

DETAILED DESCRIPTION:
In this study participants who are due to undergo elective major surgery and have an arterial line as part of their standard care will be invited to have the additional monitoring device (HDA) included as part of their care. Agreeing participants will have demographic, contact and medical history information necessary to conduct the study recorded, including a record of their intraoperative arterial line measurements.

After completing the consent process participants will receive intraoperative monitoring with Hypotension Decision Assist in addition to their standard care. The HDA monitor will be attached to the patient vital signs monitor, which will in turn be attached to the blood pressure transducer. All sampled arterial line data collected by the patient vital signs monitored will be automatically transmitted in real time to the HDA device via a serial cable attached to a digital export port of the vital signs monitor. HDA will process this input data to display, in graphical and numeric format, vital signs data and physiological parameters derived from the arterial wave form data including: Mean Arterial Pressure (MAP), systolic and diastolic blood pressure, heart rate and changes in heart rate, cardiac output and systemic vascular resistance.

The output from the study will be compared to the primary and secondary outcomes to evaluate the performance and safety of the device and to evaluate whether HDA improves control of the cardiovascular system from the anaesthetists' perspective.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) due to undergo elective surgery who are likely to have an arterial line sited as part of their standard intraoperative care.
* Recruitment after booking for surgery with sufficient time to read, understand and question study patient information prior to attending for surgery.
* Ability and willingness to provide informed consent
* Expected duration of anaesthesia > 60 minutes
* Intra-arterial monitoring is part of routine clinical care

Exclusion Criteria:

* Inability to provide informed consent
* No arterial line planned as part of their intraoperative care
* Aged < 18 years of age
* Patients with aortic regurgitation
* Patients fitted with an intra-aortic balloon pump (IABP)
* No other intra-arterial pressure management system in use
* Concurrent participation in another experimental intervention or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Display of trends in mean arterial pressure measured in millimetres of mercury (mmHg) | Intraoperative
  Operative time were HDA derives and displays mean arterial pressure (mmHg) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends in systolic blood pressure measured in millimetres of mercury (mmHg) | Intraoperative
  Operative time were HDA derives and displays systolic blood pressure (mmHg) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends in diastolic blood pressure measured in millimetres of mercury (mmHg) | Intraoperative
  Operative time were HDA derives and displays diastolic blood pressure (mmHg) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends in heart rate measured in beats per minute (bpm) | Intraoperative
  Operative time were HDA derives and displays heart rate (bpm) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends of changes in heart rate (percentage) over the previous five minutes measured as a percentage | Intraoperative
  Operative time were HDA derives and displays changes in heart rate (percentage) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends of changes in cardiac output (percentage) over the previous five minutes measured as a percentage | Intraoperative
  Operative time were HDA derives and displays changes in cardiac output (percentage) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Display of trends of changes in systemic vascular resistance (percentage) over the previous five minutes measured as a percentage | Intraoperative
  Operative time were HDA derives and displays changes in systemic vascular resistance (percentage) data that is relevant to the management of the blood pressure, hemodynamic stability and the cardiovascular system of the patient.
Adverse events (AEs) related to blood pressure attributable to HDA | Intraoperative
  Incidence, severity and causality of all AEs with delineation of those that are attributable to the use of HDA

SECONDARY OUTCOMES:
Measurement of intraoperative hypotension | Intraoperative
  Measured incidence of Mean Arterial Pressure < 65 for at least 1 minute
Number and type of intervention made by anaesthetists | Intraoperative
  Quantification of interventions related to patient cardiovascular management including fluid administered, cardiovascular active drugs administered and or drug infusion rate changes if applicable
Comparison of HDA projected trend feature | Intraoperative
  Comparison of the estimated MAP at +2mins by projected trend feature versus the observed Mean Arterial Pressure at that time as it arises.
Anaesthetists evaluation of use against a five point Likert-type scale | Intraoperative
  Anaesthetists evaluation of the ease of use and usefulness of HDA ranked in accordance with a five-point Likert-type rating scale where the minimum value is 1 (strongly disagree that HDA is useful or easy to use) and the maximum is 5 (strongly agree that HDA is useful or easy to use) .

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clutton-Brock, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Queen Elizabeth Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No